CLINICAL TRIAL: NCT05376254
Title: Three-Dimensional Assessment of Right Ventricular Function in Patients Undergoing Left Ventricular Assist Device Implantation
Brief Title: 3D Assessment of RV Function in Patients Undergoing LVAD Implantation
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00112239
Record Dates: First submitted 2022-01-27; First posted 2022-05-17 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: Right Ventricular Function; Left Ventricular Assist Device; 3D transesophageal echocardiography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This goal of this study is to analyze images of the right ventricle taken via 3D transesophageal echocardiography (TEE) during left ventricular assist device (LVAD) implantation.

DETAILED DESCRIPTION:
There are two chambers in the heart known as ventricles which are responsible for pumping blood to both the lungs and the rest of the body. The right ventricle pumps blood to the lungs for oxygenation. The left ventricle then delivers this oxygenated blood to the organs in the body. When the left ventricle is damaged enough that it is not able to effectively pump blood then it may be necessary to assist it with a mechanical pump. This pump is called left ventricular assist device (LVAD).

Left ventricular assist devices (LVADs) improve quality of life and survival in patients with end stage heart failure. However, right ventricular (RV) failure is common in 20-50% of LVAD recipients and is associated with perioperative complications.

Traditional two-dimensional ultrasound views of the right ventricle may not accurately depict how well or poorly the right ventricle is working. Three-dimensional (3D) images can overcome the limitations of two-dimensional images and are becoming more commonplace. This goal of this study is to analyze images of the right ventricle taken via 3D transesophageal echocardiography (TEE) during the LVAD implantation to help predict which patients are at higher risk of right ventricular failure within 14 days of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible to be included in the study if they receive either a left-sided:

  1. HeartMate III (Thoratec, Pleasanton, CA)
  2. HeartWare HVAD (HeartWare, Oakville CA)
  3. Levitronix CentriMag (Levitronix LLC, Waltham, MA) LVAD.

Exclusion Criteria:

* Patients will be excluded if::

  1. hemodynamic data needed to calculate PAPi or comprehensive echocardiographic images are missing
  2. additional procedures affecting cardiac geometry and/or hemodynamic measurements, such as tricuspid, mitral, and/or aortic valve repair/replacement, were performed at the time of LVAD implantation
  3. sternal closure at the end of the procedure is not possible
  4. RV mechanical support was introduced concurrently with LVAD implantation
  5. inadequate image quality required to obtain a 3D protocol
  6. known contraindication to TEE
  7. unexpected inability to advance probe into the mid-esophagus

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients coming for left ventricular assist device implantation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2027-01-19 (Estimated); Study Completion 2027-01-19 (Estimated)

PRIMARY OUTCOMES:
Left ventricular strain | 24 hours
  Prognostic indicator of hypertensive heart failure
Right ventricular fractional area of change | 24 hours
  Percentage change in the RV chamber area between end-diastole to end-systole
Right ventricular free wall strain | 24 hours
  Prognostic indicator of pulmonary arterial hypertension
Right ventricular end diastolic volume | 24 hours
  Amount of blood in the heart's right ventricle just before the heart contracts
Light ventricular end diastolic volume | 24 hours
  Amount of blood in the heart's left ventricle just before the heart contracts
Right ventricular end systolic volume | 24 hours
  Amount of blood in the heart's right ventricle just after the heart contracts
Left ventricular end systolic volume | 24 hours
  Amount of blood in the heart's left ventricle just after the heart contracts
Right ventricular ejection fraction | 24 hours
  Amount of blood being pumped out of the right ventricle each time it contracts.
Left ventricular ejection fraction | 24 hours
  Amount of blood being pumped out of the left ventricle each time it contracts.
Tricuspid annular plane systolic excursion | 24 hours
  Parameter of global right ventricular function

SECONDARY OUTCOMES:
Age | 1 day
  Demographic measure
Gender | 1 day
  Demographic measure
Body Surface Area | 1 day
  Demographic measure
Central venous pressure | 14 days
  Pressure in the thoracic vena cava near the right atrium
Pulmonary artery pulsatility index | 14 days
  Hemodynamic index
Need for right ventricular mechanical support | 14 days
  Circulatory support
Need for pulmonary vasodilators | 14 days
  Supportive medication
Need for vasopressors | 14 days
  Supportive medications
Aspartate aminotransferase | 14 days
  Lab test (> or qual to 80 IU/L)
Bilirubin | 14 days
  Lab test (> 2.0 mg/dL)
Creatinine | 14 days
  Lab test (> or equal to 2.3 mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Surita Sidhu, MD, Principal Investigator — University of Alberta
Locations (1):
- Mazankowski Alberta Heart Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Towheed A, Sabbagh E, Gupta R, Assiri S, Chowdhury MA, Moukarbel GV, Khuder SA, Schwann TA, Bonnell MR, Cooper CJ, Khouri S. Right Ventricular Dysfunction and Short-Term Outcomes Following Left-Sided Valvular Surgery: An Echocardiographic Study. J Am Heart Assoc. 2021 Feb 16;10(4):e016283. doi: 10.1161/JAHA.120.016283. Epub 2021 Feb 9. PMID 33559474
- [Background] Amzulescu MS, De Craene M, Langet H, Pasquet A, Vancraeynest D, Pouleur AC, Vanoverschelde JL, Gerber BL. Myocardial strain imaging: review of general principles, validation, and sources of discrepancies. Eur Heart J Cardiovasc Imaging. 2019 Jun 1;20(6):605-619. doi: 10.1093/ehjci/jez041. PMID 30903139
- [Background] Friedberg MK, Redington AN. Right versus left ventricular failure: differences, similarities, and interactions. Circulation. 2014 Mar 4;129(9):1033-44. doi: 10.1161/CIRCULATIONAHA.113.001375. No abstract available. PMID 24589696
- [Background] Amsallem M, Mercier O, Kobayashi Y, Moneghetti K, Haddad F. Forgotten No More: A Focused Update on the Right Ventricle in Cardiovascular Disease. JACC Heart Fail. 2018 Nov;6(11):891-903. doi: 10.1016/j.jchf.2018.05.022. Epub 2018 Oct 10. PMID 30316939
- [Background] Konstam MA, Kiernan MS, Bernstein D, Bozkurt B, Jacob M, Kapur NK, Kociol RD, Lewis EF, Mehra MR, Pagani FD, Raval AN, Ward C; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular Disease in the Young; and Council on Cardiovascular Surgery and Anesthesia. Evaluation and Management of Right-Sided Heart Failure: A Scientific Statement From the American Heart Association. Circulation. 2018 May 15;137(20):e578-e622. doi: 10.1161/CIR.0000000000000560. Epub 2018 Apr 12. PMID 29650544
- [Background] Costanzo MR, Dipchand A, Starling R, Anderson A, Chan M, Desai S, Fedson S, Fisher P, Gonzales-Stawinski G, Martinelli L, McGiffin D, Smith J, Taylor D, Meiser B, Webber S, Baran D, Carboni M, Dengler T, Feldman D, Frigerio M, Kfoury A, Kim D, Kobashigawa J, Shullo M, Stehlik J, Teuteberg J, Uber P, Zuckermann A, Hunt S, Burch M, Bhat G, Canter C, Chinnock R, Crespo-Leiro M, Delgado R, Dobbels F, Grady K, Kao W, Lamour J, Parry G, Patel J, Pini D, Towbin J, Wolfel G, Delgado D, Eisen H, Goldberg L, Hosenpud J, Johnson M, Keogh A, Lewis C, O'Connell J, Rogers J, Ross H, Russell S, Vanhaecke J; International Society of Heart and Lung Transplantation Guidelines. The International Society of Heart and Lung Transplantation Guidelines for the care of heart transplant recipients. J Heart Lung Transplant. 2010 Aug;29(8):914-56. doi: 10.1016/j.healun.2010.05.034. No abstract available. PMID 20643330
- [Background] Magunia H, Dietrich C, Langer HF, Schibilsky D, Schlensak C, Rosenberger P, Nowak-Machen M. 3D echocardiography derived right ventricular function is associated with right ventricular failure and mid-term survival after left ventricular assist device implantation. Int J Cardiol. 2018 Dec 1;272:348-355. doi: 10.1016/j.ijcard.2018.06.026. Epub 2018 Jun 8. PMID 29903518
- [Background] Haddad F, Doyle R, Murphy DJ, Hunt SA. Right ventricular function in cardiovascular disease, part II: pathophysiology, clinical importance, and management of right ventricular failure. Circulation. 2008 Apr 1;117(13):1717-31. doi: 10.1161/CIRCULATIONAHA.107.653584. No abstract available. PMID 18378625
- [Background] Lella LK, Sales VL, Goldsmith Y, Chan J, Iskandir M, Gulkarov I, Tortolani A, Brener SJ, Sacchi TJ, Heitner JF. Reduced Right Ventricular Function Predicts Long-Term Cardiac Re-Hospitalization after Cardiac Surgery. PLoS One. 2015 Jul 21;10(7):e0132808. doi: 10.1371/journal.pone.0132808. eCollection 2015. PMID 26197273
- [Background] Nagata Y, Wu VC, Kado Y, Otani K, Lin FC, Otsuji Y, Negishi K, Takeuchi M. Prognostic Value of Right Ventricular Ejection Fraction Assessed by Transthoracic 3D Echocardiography. Circ Cardiovasc Imaging. 2017 Feb;10(2):e005384. doi: 10.1161/CIRCIMAGING.116.005384. PMID 28174197
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Schneider M, Binder T. Echocardiographic evaluation of the right heart. Wien Klin Wochenschr. 2018 Jul;130(13-14):413-420. doi: 10.1007/s00508-018-1330-3. Epub 2018 Mar 19. PMID 29556779
- [Background] Mogelvang J, Stubgaard M, Thomsen C, Henriksen O. Evaluation of right ventricular volumes measured by magnetic resonance imaging. Eur Heart J. 1988 May;9(5):529-33. doi: 10.1093/oxfordjournals.eurheartj.a062539. PMID 3402468
- [Background] Dragulescu A, Grosse-Wortmann L, Fackoury C, Mertens L. Echocardiographic assessment of right ventricular volumes: a comparison of different techniques in children after surgical repair of tetralogy of Fallot. Eur Heart J Cardiovasc Imaging. 2012 Jul;13(7):596-604. doi: 10.1093/ejechocard/jer278. Epub 2011 Dec 22. PMID 22194094
- [Background] Niemann PS, Pinho L, Balbach T, Galuschky C, Blankenhagen M, Silberbach M, Broberg C, Jerosch-Herold M, Sahn DJ. Anatomically oriented right ventricular volume measurements with dynamic three-dimensional echocardiography validated by 3-Tesla magnetic resonance imaging. J Am Coll Cardiol. 2007 Oct 23;50(17):1668-76. doi: 10.1016/j.jacc.2007.07.031. PMID 17950149
- [Background] Otani K, Nabeshima Y, Kitano T, Takeuchi M. Accuracy of fully automated right ventricular quantification software with 3D echocardiography: direct comparison with cardiac magnetic resonance and semi-automated quantification software. Eur Heart J Cardiovasc Imaging. 2020 Jul 1;21(7):787-795. doi: 10.1093/ehjci/jez236. PMID 31549722
- [Background] Shimada YJ, Shiota M, Siegel RJ, Shiota T. Accuracy of right ventricular volumes and function determined by three-dimensional echocardiography in comparison with magnetic resonance imaging: a meta-analysis study. J Am Soc Echocardiogr. 2010 Sep;23(9):943-53. doi: 10.1016/j.echo.2010.06.029. PMID 20797527
- [Background] Lu MJ, Zhong WH, Liu YX, Miao HZ, Li YC, Ji MH. Sample Size for Assessing Agreement between Two Methods of Measurement by Bland-Altman Method. Int J Biostat. 2016 Nov 1;12(2):/j/ijb.2016.12.issue-2/ijb-2015-0039/ijb-2015-0039.xml. doi: 10.1515/ijb-2015-0039. PMID 27838682
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Kim J, Cohen SB, Atalay MK, Maslow AD, Poppas A. Quantitative Assessment of Right Ventricular Volumes and Ejection Fraction in Patients with Left Ventricular Systolic Dysfunction by Real Time Three-Dimensional Echocardiography versus Cardiac Magnetic Resonance Imaging. Echocardiography. 2015 May;32(5):805-12. doi: 10.1111/echo.12715. Epub 2014 Aug 11. PMID 25109323
- [Background] Leibundgut G, Rohner A, Grize L, Bernheim A, Kessel-Schaefer A, Bremerich J, Zellweger M, Buser P, Handke M. Dynamic assessment of right ventricular volumes and function by real-time three-dimensional echocardiography: a comparison study with magnetic resonance imaging in 100 adult patients. J Am Soc Echocardiogr. 2010 Feb;23(2):116-26. doi: 10.1016/j.echo.2009.11.016. PMID 20152692
- [Background] van der Zwaan HB, Helbing WA, McGhie JS, Geleijnse ML, Luijnenburg SE, Roos-Hesselink JW, Meijboom FJ. Clinical value of real-time three-dimensional echocardiography for right ventricular quantification in congenital heart disease: validation with cardiac magnetic resonance imaging. J Am Soc Echocardiogr. 2010 Feb;23(2):134-40. doi: 10.1016/j.echo.2009.12.001. PMID 20152693
- [Background] Medvedofsky D, Addetia K, Patel AR, Sedlmeier A, Baumann R, Mor-Avi V, Lang RM. Novel Approach to Three-Dimensional Echocardiographic Quantification of Right Ventricular Volumes and Function from Focused Views. J Am Soc Echocardiogr. 2015 Oct;28(10):1222-31. doi: 10.1016/j.echo.2015.06.013. Epub 2015 Aug 1. PMID 26237996